CLINICAL TRIAL: NCT00390806
Title: A Randomized, Phase III, Open-Label Study of Oral Topotecan Plus Whole-Brain Radiation Therapy (WBRT) Compared With WBRT Alone in Patients With Brain Metastases From Non-Small Cell Lung Cancer
Brief Title: Oral HYCAMTIN Plus Whole Brain Radiation Therapy In Treatment Of Brain Metastases Resulting From Non-Small Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HYT105962
Record Dates: First submitted 2006-10-19; First posted 2006-10-20 (Estimated); Results first posted 2014-01-20 (Estimated); Last update posted 2014-01-20 (Estimated); Status verified 2013-12

CONDITIONS: Lung Cancer, Non-Small Cell
Keywords: Brain metastases from Non-Small Cell Lung Cancer; Brain metastases brain tumor lung cancer oral chemotherapy HYCAMTIN topotecan NSCLC WBRT whole brain radiation
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Topotecan; Capsules; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- topotecan plus radiation (Experimental): topotecan 1.1 mg/m2 followed by whole brain radiation 3 Gy/day for 10 days, followed by optional continuation therapy with topotecan 2.3 mg/m2 for 5 days Q21 days as monotherapy.
  Interventions: Drug: HYCAMTIN, oral capsules; Radiation: Radiation
- Whole brain radiation (Active Comparator): Whole brain radiation 3 Gy/day for 10 days
  Interventions: Radiation: Radiation

INTERVENTIONS:
Drug: HYCAMTIN, oral capsules — topotecan oral capsules 1.1 mg/m2
  Other Names: HYCAMTIN; oral capsules
  Arms: topotecan plus radiation
Radiation: Radiation — Whole brain radiation

SUMMARY:
The current prognosis for patients with metastatic brain cancer from NSCLC is very poor. The current standard treatment for this disease is radiation therapy to the brain. The goal of the current study is to test whether the combination of orally administered HYCAMTIN capsules and whole brain radiation therapy will prolong the survival time of patients with this potentially serious condition.

ELIGIBILITY:
Inclusion criteria:

* At least one measurable cancerous lesion in the brain from primary non-small cell lung cancer (NSCLC)
* Must have received previous chemotherapy
* Must be 18 years of age of greater
* Must be Easter Cooperative Oncology Group (ECOG) Performance Status 0, 1, 2
* At least 2 weeks must have elapsed since any surgery
* At least 4 weeks must have elapsed since any radiation to a non-CNS site
* Must have adequate bone marrow, renal, and live capacities
* Women must be of non-childbearing potential or practice adequate birth control
* Males must practice adequate methods of birth control
* Must sign written informed consent

Exclusion criteria:

* Previous whole brain radiation therapy
* Prior treatment with topotecan
* Investigational agent within 30 days or 5 half-live
* Concomitant therapy with inhibitors of breast cancer resistance protein (BCRP) or P-glycoprotein such as erlotinib or gefitinib
* Primary or secondary immunodeficiencies
* Gastrointestinal conditions that affect GI absorption or motility
* Uncontrolled emesis
* Brain metastasis at time of initial diagnosis of NSCLC
* History of other malignancy except in situ carcinoma of cervix; nonmelanomatous skin cancer, low grade prostate cancer
* Pregnant or intending to become pregnant or intending to father a baby
* Any severe concurrent medical condition that could affect compliance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 472 (Actual)
Dates: Start 2006-12; Primary Completion 2012-07 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (79):
- United States (43):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Glendale, Arizona
  - GSK Investigational Site, Hot Springs, Arkansas
  - GSK Investigational Site, Anaheim, California
  - GSK Investigational Site, Duarte, California
  - GSK Investigational Site, Pleasant Hill, California
  - GSK Investigational Site, Aurora, Colorado
  - GSK Investigational Site, Lakeland, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Elk Grove Village, Illinois
  - GSK Investigational Site, Galesburg, Illinois
  - GSK Investigational Site, Park Ridge, Illinois
  - GSK Investigational Site, Rockford, Illinois
  - GSK Investigational Site, Skokie, Illinois
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Westwood, Kansas
  - GSK Investigational Site, Paducah, Kentucky
  - GSK Investigational Site, Metairie, Louisiana
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, Jackson, Mississippi
  - GSK Investigational Site, Columbia, Missouri
  - GSK Investigational Site, Kansas City, Missouri
  - GSK Investigational Site, Lincoln, Nebraska
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Albuquerque, New Mexico
  - GSK Investigational Site, Albany, New York
  - GSK Investigational Site, Buffalo, New York
  - GSK Investigational Site, The Bronx, New York
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Eugene, Oregon
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Bedford, Texas
  - GSK Investigational Site, Corpus Christi, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Duncanville, Texas
  - GSK Investigational Site, Fort Worth, Texas
  - GSK Investigational Site, Lubbock, Texas
  - GSK Investigational Site, Sherman, Texas
  - GSK Investigational Site, Sugarland, Texas
  - GSK Investigational Site, Everett, Washington
  - GSK Investigational Site, Vancouver, Washington
  - GSK Investigational Site, Madison, Wisconsin
- Canada (9):
  - GSK Investigational Site, Moncton, New Brunswick
  - GSK Investigational Site, Hamilton, Ontario
  - GSK Investigational Site, Kingston, Ontario
  - GSK Investigational Site, London, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Greenfield Park, Quebec
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Québec, Quebec
  - GSK Investigational Site, Sherbrooke, Quebec
- Hungary (12):
  - GSK Investigational Site, Budapest
  - GSK Investigational Site, Csorna
  - GSK Investigational Site, Győr
  - GSK Investigational Site, Gyula
  - GSK Investigational Site, Mátraháza
  - GSK Investigational Site, Miskolc
  - GSK Investigational Site, Nyíregyháza
  - GSK Investigational Site, Pécs
  - GSK Investigational Site, Székesfehérvár
  - GSK Investigational Site, Szombathely
  - GSK Investigational Site, Törökbálint
  - GSK Investigational Site, Zalaegerszeg-Pozva
- Poland (6):
  - GSK Investigational Site, Bialystok
  - GSK Investigational Site, Bydgoszcz
  - GSK Investigational Site, Gdansk
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Olsztyn
  - GSK Investigational Site, Poznan
- Russia (6):
  - GSK Investigational Site, Kazan'
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Obninsk
  - GSK Investigational Site, Orenburg
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Voronezh
- Slovakia (3):
  - GSK Investigational Site, Banská Bystrica
  - GSK Investigational Site, Bratislava
  - GSK Investigational Site, Nitra

RESULTS

PARTICIPANT FLOW:
Groups:
- Chemoradiation: Topotecan Plus WBRT: Participants received topotecan 1.1 milligrams per meters squared per day (mg/m2/day), orally followed approximately 2 hours later by whole-brain radiation therapy (WBRT) 3 Gray (Gy)/day to midline over the course of 10 days. After a 2-week washout period, participants completing chemoradiation and willing to participate in the Continuation Phase of the study received oral topotecan 2.3 mg/m2/day for 5 days, every 21 days, as monotherapy provided the baseline hematologic requirements were met. Monotherapy continued until disease progression or discontinuation. Chemoradiation participants choosing not to participate in the Continuation Phase may have received other chemotherapies or best supportive care, as determined by the investigator.
- Radiation: WBRT Alone: Participants received WBRT 3 Gy/day for 10 days. Participants may have received other chemotherapies or best supportive care, as determined by the investigator.
Period: Overall Study
Arm/Group | Chemoradiation: Topotecan Plus WBRT | Radiation: WBRT Alone
Started | 236 | 236
Ongoing | 4 | 2
Completed | 206 | 204
Not Completed | 30 | 32
Not completed — Lost to Follow-up | 7 | 6
Not completed — Protocol Violation | 2 | 2
Not completed — Withdrawal by Subject | 12 | 15
Not completed — Investigator Decision | 4 | 6
Not completed — Death | 1 | 0
Not completed — Physician Decision | 0 | 1
Not completed — Ongoing | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Chemoradiation: Topotecan Plus WBRT | Radiation: WBRT Alone | Total
Number analyzed (Participants) | 236 | 236 | 472
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.4 (8.56) | 57.8 (8.65) | 58.6 (8.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 84 | 78 | 162
  Male | 152 | 158 | 310
Race/Ethnicity, Customized [Number; unit: participants]
  African American/African Heritage (Her.) | 3 | 1 | 4
  Central/South Asian Heritage | 1 | 0 | 1
  Japanese/East Asian Heritage/South East Asian Her. | 0 | 3 | 3
  Native Hawaiian or other Pacific Islander | 1 | 0 | 1
  White | 230 | 232 | 462
  Asian & White | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Overall survival is defined as the time from randomization until the date of death due to any cause. The date of last contact was used for those participants who had not died or were lost to follow-up. These participants were classified as having been censored.
Time Frame: From the time of Randomization until the date of death due to any cause (up to 195 weeks)
Population: Intent-to-Treat (ITT) Population: all randomized participants. Participants were analyzed by the treatment to which they were randomized, even if this differed from the treatment they actually received.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Chemoradiation: Topotecan Plus WBRT | Radiation: WBRT Alone
Number analyzed (Participants) | 236 | 236
months | 4.0 [3.4 to 4.8] | 3.6 [3.0 to 4.0]
Statistical Analysis 1: Comparison: Chemoradiation: Topotecan Plus WBRT vs Radiation: WBRT Alone; Test type: Superiority or Other; p = 0.1862, Log Rank — p-value from a stratified log-rank test is adjusted for Recursive Partitioning Analysis (RPA) class and the number of brain lesions at Screening; Hazard Ratio (HR) = 0.88, 95% CI 2-sided [0.73 to 1.07] — The hazard ratio is estimated using a Pike estimator. The hazard ratio from a stratified log-rank test is adjusted for RPA class and the number of brain lesions at Screening

2. Secondary Outcome: Six-month Survival
Description: Six-month survival is defined as the percentage of participants alive at 6 months following randomization. The date of last contact was used for those participants who had not died or were lost to follow-up. These participants were classified as having been censored.
Time Frame: Month 6
Population: ITT Population
Measure: Number; unit: percentage of participants
Arm/Group | Chemoradiation: Topotecan Plus WBRT | Radiation: WBRT Alone
Number analyzed (Participants) | 236 | 236
percentage of participants | 36 | 28

3. Secondary Outcome: Number of Participants With a Complete Response (CR) or a Partial Response (PR) (Central Nervous System [CNS]-Radiologic)
Description: The number of participants achieving either a CR or PR, per World Health Organization (WHO) Criteria, in the CNS was assessed. CR is defined as the complete disappearance of all known measurable (Must be accurately measured in >=1 dimension) and nonmeasurable disease, without clinical, laboratory, or radiological evidence of recurrence for at least 4 weeks. CR may have been defined in participants with measurable and/or non-measurable disease at Screening. PR is defined as at least a 50% decrease in the sum of the products of the greatest length and perpendicular width of all measurable disease with no clear increase in nonmeasurable disease in participants without measurable disease. In both cases, there must have been no appearance of new disease, and no clinical, laboratory, or radiological evidence of disease progression for at least 4 weeks. Assessment of response was performed by the investigator and was based on unconfirmed responses.
Time Frame: From the time of Randomization until the time of CR or PR (up to 75 weeks)
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Chemoradiation: Topotecan Plus WBRT | Radiation: WBRT Alone
Number analyzed (Participants) | 236 | 236
participants
  Complete response | 23 | 11
  Partial response | 63 | 61

4. Secondary Outcome: Time to Response (TTR) (CNS-radiologic)
Description: TTR is defined as the time from Randomization until the first documented evidence of CR or PR in the CNS. CR is defined as the complete disappearance of all known measurable (Must be accurately measured in >=1 dimension) and nonmeasurable disease, without clinical, laboratory, or radiological evidence of recurrence for at least 4 weeks. CR may have been defined in participants with measurable and/or non-measurable disease at Screening. PR is defined as at least a 50% decrease in the sum of the products of the greatest length and perpendicular width of all measurable disease with no clear increase in nonmeasurable disease in participants without measurable disease. In both cases, there must have been no appearance of new disease, and no clinical, laboratory, or radiological evidence of disease progression for at least 4 weeks. Assessment of response was performed by the investigator and was based on unconfirmed responses.
Time Frame: From the time of Randomization until the first documented evidence of CR or PR (up to 75 weeks)
Population: ITT Population. Only those participants with a CR, PR, or a missing response were assessed. TTR was analyzed with censoring for extended loss to follow-up to account for two or more missed response assessments before a TTR event. The date of the last adequate CNS assessment before extended loss to follow-up was used for censored participants.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Chemoradiation: Topotecan Plus WBRT | Radiation: WBRT Alone
Number analyzed (Participants) | 173 | 170
weeks | 8.0 [7.7 to 8.1] | 8.1 [6.0 to 8.1]

5. Secondary Outcome: Time to Progression (TTP) (CNS-radiologic)
Description: TTP is defined as the time from Randomization until the first documented sign of disease progression in the CNS. Progressive disease (PD) is defined as an increase >=25% in any measurable lesion or, in participants with non-measurable disease only, an estimation of an increase >=25%. In both cases, determination of progression included the appearance of any new lesions, or signification worsening of conditions presumed to be related to malignancy. Participants with clinical or laboratory evidence of possible disease progression were to be evaluated radiologically. TTP was analyzed with censoring for extended loss to follow-up to account for two or more missed assessments before a TTP event. The date of the last adequate CNS assessment before extended loss to follow-up was used for censored participants.
Time Frame: From the time of Randomization until the first documented sign of disease progression (up to 75 weeks)
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Chemoradiation: Topotecan Plus WBRT | Radiation: WBRT Alone
Number analyzed (Participants) | 236 | 236
weeks | 9.7 [8.1 to 13.9] | 9.7 [8.3 to 10.9]

6. Secondary Outcome: Time to Progression (TTP) (All Sites of Disease-radiologic)
Description: TTP is defined as the time from Randomization until the first documented sign of disease progression in all sites of disease. Progressive disease (PD) is defined as an increase >=25% in any measurable lesion or, in participants with non-measurable disease only, an estimation of an increase >=25%. In both cases, determination of progression included the appearance of any new lesions, or signification worsening of conditions presumed to be related to malignancy. Participants with clinical or laboratory evidence of possible disease progression were to be evaluated radiologically. TTP was analyzed with censoring for extended loss to follow-up to account for two or more missed assessments before a TTP event. The date of the last adequate CNS assessment before extended loss to follow-up was used for censored participants.
Time Frame: From the time of Randomization until the first documented sign of disease progression (up to 75 weeks)
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Chemoradiation: Topotecan Plus WBRT | Radiation: WBRT Alone
Number analyzed (Participants) | 236 | 236
weeks | 8.0 [6.7 to 8.7] | 7.7 [6.1 to 8.1]

7. Secondary Outcome: Number of Participants Who Ranked Each Individual Indicated Neurological Sign and Symptom as None, Mild, Moderate, or Severe at Months 1 and 3
Description: Neurological signs and symptoms data were derived from a participant-reported diary. The participants were asked to assess the following signs and symptoms on a scale of none, mild, moderate, or severe at Months 1 and 3: headache, problems with balance/coordination (PB/C), leg weakness, arm weakness, loss of feeling/numbness (LofF/N), speech difficulty (SD), confusion, loss of memory (LofM), drowsiness, nausea, vomiting, dizziness, visual problems (VP), seizures, leg/ankle swelling (L/AS), heart burn, difficulty sleeping (DS), tiredness, and appetite/weight gain (A/WG).
Time Frame: Months 1 and 3
Population: ITT Population. Only those participants who were assessed for the indicated sign and symptom at the indicated time point were analyzed.
Measure: Number; unit: participants
Arm/Group | Chemoradiation: Topotecan Plus WBRT | Radiation: WBRT Alone
Number analyzed (Participants) | 179 | 189
participants
  Headache, Month 1, none, n=179, 189 | 93 | 106
  Headache, Month 1, mild, n=179, 189 | 71 | 68
  Headache, Month 1, moderate, 179, 189 | 11 | 13
  Headache, Month 1, severe, 179, 189 | 4 | 2
  Headache, Month 3, none, n=109, 111 | 69 | 53
  Headache, Month 3, mild, n=109, 111 | 33 | 41
  Headache, Month 3, moderate, n=109, 111 | 5 | 14
  Headache, Month 3, severe, n=109, 111 | 2 | 3
  PB/C, Month 1, none, n=179, 188 | 84 | 79
  PB/C, Month 1, mild, n=179, 188 | 66 | 71
  PB/C, Month 1, moderate, n=179, 188 | 22 | 30
  PB/C, Month 1, severe, n=179, 188 | 7 | 8
  PB/C, Month 3, none, n=109, 111 | 69 | 46
  PB/C, Month 3, mild, n=109, 111 | 28 | 36
  PB/C, Month 3, moderate, n=109, 111 | 10 | 18
  PB/C, Month 3, severe, n=109, 111 | 2 | 11
  Leg weakness, Month 1, none, n=179, 188 | 47 | 59
  Leg weakness, Month 1, mild, n=179, 188 | 73 | 72
  Leg weakness, Month 1, moderate, n=179, 188 | 41 | 41
  Leg weakness, Month 1, severe, n=179, 188 | 18 | 16
  Leg weakness, Month 3, none, n=109, 111 | 28 | 34
  Leg weakness, Month 3, mild, n=109, 111 | 51 | 37
  Leg weakness, Month 3, moderate, n=109, 111 | 20 | 19
  Leg weakness, Month 3, severe, n=109, 111 | 10 | 21
  Arm weakness, Month 1, none, n=179, 188 | 96 | 97
  Arm weakness, Month 1, mild, n=179, 188 | 55 | 60
  Arm weakness, Month 1, moderate, n=179, 188 | 23 | 18
  Arm weakness, Month 1, severe, n=179, 188 | 5 | 13
  Arm weakness, Month 3, none, n=109, 111 | 60 | 53
  Arm weakness, Month 3, mild, n=109, 111 | 39 | 34
  Arm weakness, Month 3, molderate, n=109, 111 | 8 | 16
  Arm weakness, Month 3, severe, n=109, 111 | 2 | 8
  LofF/N, Month 1, none, n=179, 188 | 101 | 11
  LofF/N, Month 1, mild, n=179, 188 | 53 | 43
  LofF/N, Month 1, moderate, n=179, 188 | 17 | 25
  LofF/N, Month 1, severe, n=179, 188 | 8 | 9
  LofF/N, Month 3, none, n=109, 111 | 73 | 66
  LofF/N, Month 3, mild, n=109, 111 | 28 | 27
  LofF/N, Month 3, moderate, n=109, 111 | 3 | 11
  LofF/N, Month 3, severe, n=109, 111 | 5 | 7
  SD, Month 1, none, n=179, 188 | 151 | 137
  SD, Month 1, mild, n=179, 188 | 16 | 40
  SD, Month 1, moderate, n=179, 188 | 9 | 9
  SD, Month 1, severe, n=179, 188 | 3 | 2
  SD, Month 3, none, n=109, 110 | 94 | 78
  SD, Month 3, mild, n=109, 110 | 11 | 22
  SD, Month 3, moderate, n=109, 110 | 2 | 8
  SD, Month 3, severe, n=109, 110 | 2 | 2
  Confusion, Month 1, none, n=179, 188 | 150 | 148
  Confusion, Month 1, mild, n=179, 188 | 20 | 32
  Confusion, Month 1, moderate, n=179, 188 | 6 | 7
  Confusion, Month 1, severe, n=179, 188 | 3 | 1
  Confusion, Month 3, none, n=109, 110 | 99 | 71
  Confusion, Month 3, mild, n=109, 110 | 7 | 29
  Confusion, Month 3, moderate, n=109, 110 | 2 | 9
  Confusion, Month 3, severe, n=109, 110 | 1 | 1
  LofM, Month 1, none, n=179, 188 | 149 | 141
  LofM, Month 1, mild, n=179, 188 | 20 | 41
  LofM, Month 1, moderate, n=179, 188 | 8 | 5
  LofM, Month 1, severe, n=179, 188 | 2 | 1
  LofM, Month 3, none, n=109, 110 | 93 | 78
  LofM, Month 3, mild, n=109, 110 | 14 | 25
  LofM, Month 3, moderate, n=109, 110 | 1 | 6
  LofM, Month 3, severe, n=109, 110 | 1 | 1
  Drowsiness, Month 1, none, n=179, 188 | 90 | 96
  Drowsiness, Month 1, mild, n=179, 188 | 55 | 59
  Drowsiness, Month 1, moderate, n=179, 188 | 25 | 26
  Drowsiness, Month 1, severe, n=179, 188 | 9 | 7
  Drowsiness, Month 3, none, n=109, 111 | 50 | 44
  Drowsiness, Month 3, mild, n=109, 111 | 42 | 40
  Drowsiness, Month 3, moderate, n=109, 111 | 15 | 15
  Drowsiness, Month 3, severe, n=109, 111 | 2 | 12
  Nausea, Month 1, none, n=179, 188 | 125 | 142
  Nausea, Month 1, mild, n=179, 188 | 38 | 36
  Nausea, Month 1, moderate, n=179, 188 | 12 | 10
  Nausea, Month 1, severe, n=179, 188 | 4 | 0
  Nausea, Month 3, none, n=109, 111 | 70 | 73
  Nausea, Month 3, mild, n=109, 111 | 31 | 29
  Nausea, Month 3, moderate, n=109, 111 | 7 | 6
  Nausea, Month 3, severe, n=109, 111 | 1 | 3
  Vomiting, Month 1, none, n=179, 188 | 153 | 164
  Vomiting, Month 1, mild, n=179, 188 | 20 | 19
  Vomiting, Month 1, moderate, n=179, 188 | 4 | 4
  Vomiting, Month 1, severe, n=179, 188 | 2 | 1
  Vomiting, Month 3, none, n=109, 111 | 89 | 91
  Vomiting, Month 3, mild, n=109, 111 | 15 | 15
  Vomiting, Month 3, moderate, n=109, 111 | 4 | 3
  Vomiting, Month 3, severe=109, 111 | 1 | 2
  Dizziness, Month 1, none, n=179, 188 | 96 | 94
  Dizziness, Month 1, mild, n=179, 188 | 58 | 70
  Dizziness, Month 1, moderate, n=179, 188 | 22 | 21
  Dizziness, Month 1, severe, n=179, 188 | 3 | 3
  Dizziness, Month 3, none, n=109, 111 | 64 | 54
  Dizziness, Month 3, mild, n=109, 111 | 35 | 36
  Dizziness, Month 3, moderate, n=109, 111 | 7 | 14
  Dizziness, Month 3, severe, n=109, 111 | 3 | 7
  VP, Month 1, none, n=179, 188 | 103 | 117
  VP, Month 1, mild, n=179, 188 | 54 | 53
  VP, Month 1, moderate, n=179, 188 | 17 | 16
  VP, Month 1, severe, n=179, 188 | 5 | 2
  VP, Month 3, none, n=109, 111 | 72 | 69
  VP, Month 3, mild, n=109, 111 | 29 | 28
  VP, Month 3, moderate, n=109, 111 | 7 | 10
  VP, Month 3, severe, n=109, 111 | 1 | 4
  Seizures, Month 1, none, n=179, 188 | 173 | 179
  Seizures, Month 1, mild, n=179, 188 | 5 | 7
  Seizures, Month 1, moderate, n=179, 188 | 1 | 2
  Seizures, Month 1, severe, n=179, 188 | 0 | 0
  Seizures, Month 3, none, n=109, 110 | 108 | 102
  Seizures, Month 3, mild, n=109, 110 | 0 | 4
  Seizures, Month 3, moderate, n=109, 110 | 1 | 3
  Seizures, Month 3, severe, n=109, 110 | 0 | 1
  L/AS, Month 1, none, n=179, 188 | 141 | 138
  L/AS, Month 1, mild, n=179, 188 | 21 | 29
  L/AS, Month 1, moderate, n=179, 188 | 12 | 15
  L/AS, Month 1, severe, n=179, 188 | 5 | 6
  L/AS, Month 3, none, n=109, 111 | 86 | 85
  L/AS, Month 3, mild, n=109, 111 | 19 | 19
  L/AS, Month 3, moderate, n=109, 111 | 3 | 6
  L/AS, Month 3, severe, n=109, 111 | 1 | 1
  Heartburn, Month 1, none, n=179, 188 | 142 | 151
  Heartburn, Month 1, mild, n=179, 188 | 26 | 27
  Heartburn, Month 1, moderate, n=179, 188 | 9 | 9
  Heartburn, Month 1, severe, n=179, 188 | 2 | 1
  Heartburn, Month 3, none, n=109, 111 | 87 | 86
  Heartburn, Month 3, mild, n=109, 111 | 16 | 18
  Heartburn, Month 3, moderate, n=109, 111 | 4 | 6
  Heartburn, Month 3, severe, n=109, 111 | 2 | 1
  DS, Month 1, none, n=179, 188 | 112 | 109
  DS, Month 1, mild, n=179, 188 | 41 | 48
  DS, Month 1, moderate, n=179, 188 | 15 | 24
  DS, Month 1, severe, n=179, 188 | 11 | 7
  DS, Month 3, none, n=109, 110 | 78 | 71
  DS, Month 3, mild, n=109, 110 | 20 | 23
  DS, Month 3, moderate, n=109, 110 | 8 | 12
  DS, Month 3, severe, n=109, 110 | 3 | 4
  Tiredness, Month 1, none, n=179, 188 | 42 | 42
  Tiredness, Month 1, mild, n=179, 188 | 75 | 85
  Tiredness, Month 1, moderate, n=179, 188 | 46 | 44
  Tiredness, Month 1, severe, n=179, 188 | 16 | 17
  Tiredness, Month 3, none, n=109, 111 | 28 | 21
  Tiredness, Month 3, mild, n=109, 111 | 52 | 42
  Tiredness, Month 3, moderate, n=109, 111 | 19 | 32
  Tiredness, Month 3, severe, n=109, 111 | 10 | 16
  A/WG, Month 1, none, n=179, 188 | 107 | 113
  A/WG, Month 1, mild, n=179, 188 | 42 | 41
  A/WG, Month 1, moderate, n=179, 188 | 19 | 29
  A/WG, Month 1, severe, n=179, 188 | 11 | 5
  A/WG, Month 3, none, n=108, 111 | 71 | 73
  A/WG, Month 3, mild, n=108, 111 | 27 | 23
  A/WG, Month 3, moderate, n=108, 111 | 4 | 11
  A/WG, Month 3, severe, n=108, 111 | 6 | 4

8. Secondary Outcome: Number of Participants With the Indicated Investigator Assessment for the Neurological Sign and Symptom of Level of Consciousness at Baseline, Month 1, and Month 3
Description: The investigator assessed participants for the neurological sign and symptom of level of consciousness and assigned each participant to one of the following categories: normal; somnolence or sedation not interfering with function (not intefering); somnolence or sedation interfering with function, but not activities of daily living (ADLs) (interfering); obtundation or stupor, difficult to arouse, inteferring with ADLs (obtundation or stupor); coma.
Time Frame: Baseline, Month 1, and Month 3
Population: ITT Population. Only those participants who were assessed at the indicated time point were analyzed. If no data are presented for a particular status at a particular time point, then no participants had that status at that time point.
Measure: Number; unit: participants
Arm/Group | Chemoradiation: Topotecan Plus WBRT | Radiation: WBRT Alone
Number analyzed (Participants) | 230 | 228
participants
  Baseline, normal, n=230, 228 | 219 | 216
  Month 1, normal, n=178, 180 | 171 | 169
  Month 3, normal, n=109, 107 | 102 | 92
  Baseline, not interfering, n=230, 228 | 7 | 9
  Month 1, not interfering, n=178, 180 | 5 | 7
  Month 3, not interfering, n=109, 107 | 3 | 8
  Baseline, interfering, n=230, 228 | 3 | 3
  Month 1, interfering, n=178, 180 | 0 | 4
  Month 3, interfering, n=109, 107 | 3 | 5
  Baseline, obtundation and stupor, n=230, 228 | 1 | 0
  Month 1, obtundation and stupor, n=178, 180 | 2 | 0
  Month 3, obtundation and stupor, n=109, 107 | 1 | 2

9. Secondary Outcome: Number of Participants With the Indicated Investigator Assessment for the Neurological Sign and Symptom of Headache at Baseline, Month 1, and Month 3
Description: The investigator (per Common Terminology Criteria for Adverse Events [CTCAE], version 3.0) assessed participants for headache and assigned each participant to one of the following categories: absent, Grade (G) 1, G 2, G 3, G 4, and G 5. Grade refers to the severity of the AE. The CTCAE displays G 1 through 5 with unique clinical descriptions of severity for each AE based on this general guideline: G 1: mild, asymptomatic or mild symptoms, clinical or diagnostic observations only, intervention not indicated; G 2: moderate, minimal, local or noninvasive intervention indicated, limiting age-appropriate instrumental ADL; G 3: severe or medically significant but not immediately life-threatening, hospitalization or prolongation of hospitalization indicated, disabling, limiting self care ADL; G 4: life-threatening consequences, urgent intervention indicated; G 5: death related to AE.
Time Frame: Baseline, Month 1, and Month 3
Population: ITT Population. Only those participants who were assessed at the indicated time point were analyzed. If no data are presented for a particular grade at a particular time point, then no participants had an event of that grade at that time point.
Measure: Number; unit: participants
Arm/Group | Chemoradiation: Topotecan Plus WBRT | Radiation: WBRT Alone
Number analyzed (Participants) | 230 | 228
participants
  Baseline, absent, n=230, 228 | 141 | 146
  Month 1, absent, n=178, 180 | 126 | 127
  Month 3, absent, n=109, 107 | 85 | 74
  Baseline, Grade 1, n=230, 228 | 62 | 55
  Month 1, Grade 1, n=178, 180 | 43 | 38
  Month 3, Grade 1, n=109, 107 | 17 | 23
  Baseline, Grade 2, n=230, 228 | 25 | 23
  Month 1, Grade 2, n=178, 180 | 9 | 14
  Month 3, Grade 2, n=109, 107 | 7 | 10
  Baseline, Grade 3, n=230, 228 | 2 | 4
  Month 1, Grade 3, n=178, 180 | 0 | 1

10. Secondary Outcome: Number of Participants With the Indicated Investigator Assessment for the Neurological Sign and Symptom of Dizziness/Lightheadedness at Baseline, Month 1, and Month 3
Description: The investigator (per CTCAE, version 3.0) assessed participants for dizziness/lightheadedness and assigned each participant to one of the following categories: absent, G 1, G 2, G 3, G 4, and G 5. Grade refers to the severity of the AE. The CTCAE displays G 1 through 5 with unique clinical descriptions of severity for each AE based on this general guideline: G 1: mild, asymptomatic or mild symptoms, clinical or diagnostic observations only, intervention not indicated; G 2: moderate, minimal, local or noninvasive intervention indicated, limiting age-appropriate instrumental ADL; G 3: severe or medically significant but not immediately life-threatening, hospitalization or prolongation of hospitalization indicated, disabling, limiting self care ADL; G 4: life-threatening consequences, urgent intervention indicated; G 5: death related to AE.
Time Frame: Baseline, Month 1, and Month 3
Population: as for outcome 9
Measure: Number; unit: participants
Arm/Group | Chemoradiation: Topotecan Plus WBRT | Radiation: WBRT Alone
Number analyzed (Participants) | 230 | 228
participants
  Baseline, absent, n=230, 228 | 160 | 151
  Month 1, absent, n=178, 180 | 124 | 128
  Month 3, absent, n=109, 107 | 76 | 76
  Baseline, Grade 1, n=230, 228 | 45 | 47
  Month 1, Grade 1, n=178, 180 | 44 | 36
  Month 3, Grade 1, n=109, 107 | 21 | 20
  Baseline, Grade 2, n=230, 228 | 21 | 26
  Month 1, Grade 2, n=178, 180 | 7 | 14
  Month 3, Grade 2, n=109, 107 | 9 | 9
  Baseline, Grade 3, n=230, 228 | 4 | 4
  Month 1, Grade 3, n=178, 180 | 3 | 2
  Month 3, Grade 3, n=109, 107 | 3 | 2

11. Secondary Outcome: Number of Participants With the Indicated Investigator Assessment for the Neurological Sign and Symptom of Vertigo at Baseline, Month 1, and Month 3
Description: The investigator (per CTCAE, version 3.0) assessed participants for vertigo and assigned each participant to one of the following categories: absent, G 1, G 2, G 3, G 4, and G 5. Grade refers to the severity of the AE. The CTCAE displays G 1 through 5 with unique clinical descriptions of severity for each AE based on this general guideline: G 1: mild, asymptomatic or mild symptoms, clinical or diagnostic observations only, intervention not indicated; G 2: moderate, minimal, local or noninvasive intervention indicated, limiting age-appropriate instrumental ADL; G 3: severe or medically significant but not immediately life-threatening, hospitalization or prolongation of hospitalization indicated, disabling, limiting self care ADL; G 4: life-threatening consequences, urgent intervention indicated; G 5: death related to AE.
Time Frame: Baseline, Month 1, and Month 3
Population: as for outcome 9
Measure: Number; unit: participants
Arm/Group | Chemoradiation: Topotecan Plus WBRT | Radiation: WBRT Alone
Number analyzed (Participants) | 230 | 228
participants
  Baseline, absent, n=230, 228 | 180 | 173
  Month 1, absent, n=178, 180 | 148 | 150
  Month 3, absent, n=109, 107 | 90 | 86
  Baseline, Grade 1, n=230, 228 | 26 | 30
  Month 1, Grade 1, n=178, 180 | 19 | 19
  Month 3, Grade 1, n=109, 107 | 14 | 13
  Baseline, Grade 2, n=230, 228 | 19 | 22
  Month 1, Grade 2, n=178, 180 | 7 | 9
  Month 3, Grade 2, n=109, 107 | 4 | 6
  Baseline, Grade 3, n=230, 228 | 5 | 3
  Month 1, Grade 3, n=178, 180 | 3 | 2
  Month 3, Grade 3, n=109, 107 | 1 | 2
  Month 1, Grade 4, n=178, 180 | 1 | 0

12. Secondary Outcome: Number of Participants With the Indicated Investigator Assessment for the Neurological Sign and Symptom of Nausea/Vomiting at Baseline, Month 1, and Month 3
Description: The investigator (per CTCAE, version 3.0) assessed participants for nausea/vomiting and assigned each participant to one of the following categories: absent, G 1, G 2, G 3, G 4, and G 5. Grade refers to the severity of the AE. The CTCAE displays G 1 through 5 with unique clinical descriptions of severity for each AE based on this general guideline: G 1: mild, asymptomatic or mild symptoms, clinical or diagnostic observations only, intervention not indicated; G 2: moderate, minimal, local or noninvasive intervention indicated, limiting age-appropriate instrumental ADL; G 3: severe or medically significant but not immediately life-threatening, hospitalization or prolongation of hospitalization indicated, disabling, limiting self care ADL; G 4: life-threatening consequences, urgent intervention indicated; G 5: death related to AE.
Time Frame: Baseline, Month 1, and Month 3
Population: as for outcome 9
Measure: Number; unit: participants
Arm/Group | Chemoradiation: Topotecan Plus WBRT | Radiation: WBRT Alone
Number analyzed (Participants) | 230 | 228
participants
  Baseline, absent, n=230, 228 | 203 | 192
  Month 1, absent, n=178, 180 | 151 | 162
  Month 3, absent, n=109, 107 | 88 | 93
  Baseline, Grade 1, n=230, 228 | 19 | 22
  Month 1, Grade 1, n=178, 180 | 20 | 15
  Month 3, Grade 1, n=109, 107 | 14 | 11
  Baseline, Grade 2, n=230, 228 | 7 | 10
  Month 1, Grade 2, n=178, 180 | 6 | 3
  Month 3, Grade 2, n=109, 107 | 6 | 3
  Baseline, Grade 3, n=230, 228 | 1 | 4
  Month 1, Grade 3, n=178, 180 | 1 | 0
  Month 3, Grade 5, n=109, 107 | 1 | 0

13. Secondary Outcome: Number of Participants With the Indicated Investigator Assessment for the Neurological Sign and Symptom of Visual Problem at Baseline, Month 1, and Month 3
Description: The investigator (per CTCAE, version 3.0) assessed participants for visual problem and assigned each participant to one of the following categories: absent, G 1, G 2, G 3, G 4, and G 5. Grade refers to the severity of the AE. The CTCAE displays G 1 through 5 with unique clinical descriptions of severity for each AE based on this general guideline: G 1: mild, asymptomatic or mild symptoms, clinical or diagnostic observations only, intervention not indicated; G 2: moderate, minimal, local or noninvasive intervention indicated, limiting age-appropriate instrumental ADL; G 3: severe or medically significant but not immediately life-threatening, hospitalization or prolongation of hospitalization indicated, disabling, limiting self care ADL; G 4: life-threatening consequences, urgent intervention indicated; G 5: death related to AE.
Time Frame: Baseline, Month 1, and Month 3
Population: as for outcome 9
Measure: Number; unit: participants
Arm/Group | Chemoradiation: Topotecan Plus WBRT | Radiation: WBRT Alone
Number analyzed (Participants) | 230 | 228
participants
  Baseline, absent, n=230, 228 | 181 | 189
  Month 1, absent, n=178, 180 | 148 | 154
  Month 3, absent, n=109, 107 | 93 | 93
  Baseline, Grade 1, n=230, 228 | 22 | 25
  Month 1, Grade 1, n=178, 180 | 16 | 19
  Month 3, Grade 1, n=109, 107 | 12 | 10
  Baseline, Grade 2, n=230, 228 | 20 | 13
  Month 1, Grade 2, n=178, 180 | 11 | 6
  Month 3, Grade 2, n=109, 107 | 4 | 3
  Baseline, Grade 3, n=230, 228 | 5 | 1
  Month 1, Grade 3, n=178, 180 | 2 | 1
  Month 3, Grade 3, n=109, 107 | 0 | 1
  Baseline, Grade 4, n=230, 228 | 2 | 0
  Month 1, Grade 4, n=178, 180 | 1 | 0

14. Secondary Outcome: Number of Participants With the Indicated Investigator Assessment for the Neurological Sign and Symptom of Seizure at Baseline, Month 1, and Month 3
Description: The investigator (per CTCAE, version 3.0) assessed participants for seizure and assigned each participant to one of the following categories: absent, G 1, G 2, G 3, G 4, and G 5. Grade refers to the severity of the AE. The CTCAE displays G 1 through 5 with unique clinical descriptions of severity for each AE based on this general guideline: G 1: mild, asymptomatic or mild symptoms, clinical or diagnostic observations only, intervention not indicated; G 2: moderate, minimal, local or noninvasive intervention indicated, limiting age-appropriate instrumental ADL; G 3: severe or medically significant but not immediately life-threatening, hospitalization or prolongation of hospitalization indicated, disabling, limiting self care ADL; G 4: life-threatening consequences, urgent intervention indicated; G 5: death related to AE.
Time Frame: Baseline, Month 1, and Month 3
Population: as for outcome 9
Measure: Number; unit: participants
Arm/Group | Chemoradiation: Topotecan Plus WBRT | Radiation: WBRT Alone
Number analyzed (Participants) | 230 | 228
participants
  Baseline, absent, n=230, 228 | 218 | 216
  Month 1, absent, n=178, 180 | 175 | 178
  Month 3, absent, n=109, 107 | 109 | 101
  Baseline, Grade 1, n=230, 228 | 4 | 6
  Month 1, Grade 1, n=178, 180 | 2 | 1
  Month 3, Grade 1, n=109, 107 | 0 | 4
  Baseline, Grade 2, n=230, 228 | 6 | 6
  Month 1, Grade 2, n=178, 180 | 1 | 1
  Month 3, Grade 2, n=109, 107 | 0 | 2
  Baseline, Grade 3, n=230, 228 | 1 | 0
  Baseline, Grade 4, n=230, 228 | 1 | 0

15. Secondary Outcome: Number of Participants With the Indicated Investigator Assessment for the Neurological Sign and Symptom of Other Neurological Symptoms at Baseline, Month 1, and Month 3
Description: The investigator (per CTCAE, version 3.0) assessed participants for other neurological symptoms and assigned each participant to one of the following categories: absent, G 1, G 2, G 3, G 4, and G 5. Grade refers to the severity of the AE. The CTCAE displays G 1 through 5 with unique clinical descriptions of severity for each AE based on this general guideline: G 1: mild, asymptomatic or mild symptoms, clinical or diagnostic observations only, intervention not indicated; G 2: moderate, minimal, local or noninvasive intervention indicated, limiting age-appropriate instrumental ADL; G 3: severe or medically significant but not immediately life-threatening, hospitalization or prolongation of hospitalization indicated, disabling, limiting self care ADL; G 4: life-threatening consequences, urgent intervention indicated; G 5: death related to AE.
Time Frame: Baseline, Month 1, and Month 3
Population: as for outcome 9
Measure: Number; unit: participants
Arm/Group | Chemoradiation: Topotecan Plus WBRT | Radiation: WBRT Alone
Number analyzed (Participants) | 229 | 228
participants
  Baseline, absent, n=229, 228 | 219 | 214
  Month 1, absent, n=177, 180 | 165 | 171
  Month 3, absent, n=109, 107 | 99 | 101
  Baseline, Grade 1, n=229, 228 | 2 | 5
  Month 1, Grade 1, n=177, 180 | 2 | 6
  Month 3, Grade 1, n=109, 107 | 6 | 5
  Baseline, Grade 2, n=229, 228 | 7 | 8
  Month 1, Grade 2, n=177, 180 | 8 | 1
  Month 3, Grade 2, n=109, 107 | 3 | 1
  Baseline, Grade 3, n=229, 228 | 1 | 1
  Month 1, Grade 3, n=177, 180 | 2 | 1
  Month 1, Grade 4, n=177, 180 | 0 | 1
  Month 3, Grade 5, n=109, 107 | 1 | 0

16. Secondary Outcome: Number of Participants With the Indicated Investigator Assessment of Cranial Nerves II-XII at Baseline, Month 1, and Month 3
Description: The investigator assessed participants' status of cranial nerves II-XII and assigned each participant to one of the following categories: normal; present, not interfering with ADLs; present, interfering with ADLs; life threatening, disabling.
Time Frame: Baseline, Month 1, and Month 3
Population: as for outcome 8
Measure: Number; unit: participants
Arm/Group | Chemoradiation: Topotecan Plus WBRT | Radiation: WBRT Alone
Number analyzed (Participants) | 229 | 225
participants
  Baseline, normal, n=229, 225 | 218 | 211
  Month 1, normal, n=177, 179 | 172 | 169
  Month 3, normal, n=109, 107 | 106 | 102
  Baseline, present, not interfering, n=229, 225 | 11 | 10
  Month 1, present, not interfering, n=177, 179 | 4 | 6
  Month 3, present, not interfering, n=109, 107 | 3 | 2
  Baseline, present, interfering, n=229, 225 | 0 | 4
  Month 1, present, interfering, n=177, 179 | 1 | 4
  Month 3, present, interfering, n=109, 107 | 0 | 3

17. Secondary Outcome: Number of Participants With the Indicated Investigator Assessment of Language (Dysphasia or Aphasia) at Baseline, Month 1, and Month 3
Description: The investigator assessed participants' status of language (dysphasia or aphasia) and assigned each participant to one of the following categories: absent; awareness of receptive or expressive aphasia, not impairing ability to communicate (not impaired); receptive or expressive dysphasia, impairing ability to communicate (impaired); inability to communicate (unable).
Time Frame: Baseline, Month 1, and Month 3
Population: as for outcome 8
Measure: Number; unit: participants
Arm/Group | Chemoradiation: Topotecan Plus WBRT | Radiation: WBRT Alone
Number analyzed (Participants) | 230 | 228
participants
  Baseline, absent, n=230, 228 | 211 | 215
  Month 1, absent, n=178, 180 | 169 | 173
  Month 3, absent, n=109, 107 | 105 | 98
  Baseline, not impaired, n=230, 228 | 15 | 10
  Month 1, not impaired, n=178, 180 | 6 | 5
  Month 3, not impaired, n=109, 107 | 3 | 7
  Baseline, impaired, n=230, 228 | 3 | 3
  Month 1, impaired, n=178, 180 | 3 | 2
  Month 3, impaired, n=109, 107 | 1 | 0
  Baseline, unable, n=230, 228 | 1 | 0
  Month 3, unable, n=109, 107 | 0 | 2

18. Secondary Outcome: Number of Participants With the Indicated Investigator Assessment of Strength (Right Upper Extremity) at Baseline, Month 1, and Month 3
Description: The investigator assessed participants' status of strength (right upper extremity) and assigned each participant to one of the following categories: normal; Grade 1, asymptomatic with weakness on physical examination; Grade 2, symptomatic and interfering with function, but not interfering with ADLs; Grade 3, symptomatic and interfering with ADLs; Grade 4: bedridden or disabling.
Time Frame: Baseline, Month 1, and Month 3
Population: as for outcome 8
Measure: Number; unit: participants
Arm/Group | Chemoradiation: Topotecan Plus WBRT | Radiation: WBRT Alone
Number analyzed (Participants) | 230 | 228
participants
  Baseline, normal, n=230, 228 | 203 | 195
  Month 1, normal, n=178, 179 | 153 | 159
  Month 3, normal, n=109, 107 | 93 | 89
  Baseline, Grade 1, n=230, 228 | 15 | 16
  Month 1, Grade 1, n=178, 179 | 13 | 12
  Month 3, Grade 1, n=109, 107 | 10 | 10
  Baseline, Grade 2, n=230, 228 | 6 | 12
  Month 1, Grade 2, n=178, 179 | 6 | 5
  Month 3, Grade 2, n=109, 107 | 4 | 5
  Baseline, Grade 3, n=230, 228 | 5 | 5
  Month 1, Grade 3, n=178, 179 | 4 | 2
  Month 3, Grade 3, n=109, 107 | 2 | 3
  Baseline, Grade 4, n=230, 228 | 1 | 0
  Month 1, Grade 4, n=178, 179 | 2 | 1

19. Secondary Outcome: Number of Participants With the Indicated Investigator Assessment of Strength (Left Upper Extremity) at Baseline, Month 1, and Month 3
Description: The investigator assessed participants' status of strength (left upper extremity) and assigned each participant to one of the following categories: normal; Grade 1, asymptomatic with weakness on physical examination; Grade 2, symptomatic and interfering with function, but not interfering with ADLs; Grade 3, symptomatic and interfering with ADLs; Grade 4: bedridden or disabling.
Time Frame: Baseline, Month 1, and Month 3
Population: as for outcome 8
Measure: Number; unit: participants
Arm/Group | Chemoradiation: Topotecan Plus WBRT | Radiation: WBRT Alone
Number analyzed (Participants) | 230 | 228
participants
  Baseline, normal, n=230, 228 | 197 | 202
  Month 1, normal, n=178, 179 | 149 | 157
  Month 3, normal, n=109, 107 | 90 | 86
  Baseline, Grade 1, n=230, 228 | 16 | 13
  Month 1, Grade 1, n=178, 179 | 16 | 13
  Month 3, Grade 1, n=109, 107 | 10 | 11
  Baseline, Grade 2, n=230, 228 | 11 | 8
  Month 1, Grade 2, n=178, 179 | 8 | 5
  Month 3, Grade 2, n=109, 107 | 6 | 5
  Baseline, Grade 3, n=230, 228 | 6 | 4
  Month 1, Grade 3, n=178, 179 | 3 | 2
  Month 3, Grade 3, n=109, 107 | 3 | 4
  Baseline, Grade 4, n=230, 228 | 0 | 1
  Month 1, Grade 4, n=178, 179 | 2 | 2
  Month 3, Grade 4, n=109, 107 | 0 | 1

20. Secondary Outcome: Number of Participants With the Indicated Investigator Assessment of Strength (Right Lower Extremity) at Baseline, Month 1, and Month 3
Description: The investigator assessed participants' status of strength (right lower extremity) and assigned each participant to one of the following categories: normal; Grade 1, asymptomatic with weakness on physical examination; Grade 2, symptomatic and interfering with function, but not interfering with ADLs; Grade 3, symptomatic and interfering with ADLs; Grade 4: bedridden or disabling.
Time Frame: Baseline, Month 1, and Month 3
Population: as for outcome 8
Measure: Number; unit: participants
Arm/Group | Chemoradiation: Topotecan Plus WBRT | Radiation: WBRT Alone
Number analyzed (Participants) | 230 | 228
participants
  Baseline, normal, n=230, 228 | 196 | 189
  Month 1, normal, n=178, 180 | 137 | 145
  Month 3, normal, n=109, 107 | 81 | 80
  Baseline, Grade 1, n=230, 228 | 20 | 19
  Month 1, Grade 1, n=178, 180 | 17 | 15
  Month 3, Grade 1, n=109, 107 | 12 | 11
  Baseline, Grade 2, n=230, 228 | 9 | 16
  Month 1, Grade 2, n=178, 180 | 11 | 19
  Month 3, Grade 2, n=109, 107 | 11 | 11
  Baseline, Grade 3, n=230, 228 | 3 | 4
  Month 1, Grade 3, n=178, 180 | 9 | 0
  Month 3, Grade 3, n=109, 107 | 4 | 3
  Baseline, Grade 4, n=230, 228 | 2 | 0
  Month 1, Grade 4, n=178, 180 | 4 | 1
  Month 3, Grade 4, n=109, 107 | 1 | 2

21. Secondary Outcome: Number of Participants With the Indicated Investigator Assessment of Strength (Left Lower Extremity) at Baseline, Month 1, and Month 3
Description: The investigator assessed participants' status of strength (left lower extremity) and assigned each participant to one of the following categories: normal; Grade 1, asymptomatic with weakness on physical examination; Grade 2, symptomatic and interfering with function, but not interfering with ADLs; Grade 3, symptomatic and interfering with ADLs; Grade 4: bedridden or disabling.
Time Frame: Baseline, Month 1, and Month 3
Population: as for outcome 8
Measure: Number; unit: participants
Arm/Group | Chemoradiation: Topotecan Plus WBRT | Radiation: WBRT Alone
Number analyzed (Participants) | 230 | 228
participants
  Baseline, normal, n=230, 228 | 182 | 190
  Month 1, normal, n=178, 179 | 128 | 143
  Month 3, normal, n=109, 107 | 76 | 73
  Baseline, Grade 1, n=230, 228 | 28 | 18
  Month 1, Grade 1, n=178, 179 | 26 | 13
  Month 3, Grade 1, n=109, 107 | 11 | 11
  Baseline, Grade 2, n=230, 228 | 15 | 15
  Month 1, Grade 2, n=178, 179 | 11 | 17
  Month 3, Grade 2, n=109, 107 | 14 | 14
  Baseline, Grade 3, n=230, 228 | 4 | 3
  Month 1, Grade 3, n=178, 179 | 10 | 4
  Month 3, Grade 3, n=109, 107 | 6 | 5
  Baseline, Grade 4, n=230, 228 | 1 | 2
  Month 1, Grade 4, n=178, 179 | 3 | 2
  Month 3, Grade 4, n=109, 107 | 2 | 4

22. Secondary Outcome: Number of Participants With the Indicated Investigator Assessment of Sensation at Baseline, Month 1, and Month 3
Description: The investigator assessed participants' status of sensation and assigned each participant to one of the following categories: normal; loss of deep tendon reflexes or paresthesia, but not interfering with function (not interfering with function); objective sensory loss or paresthesia interfering with function, but not interfering with ADLs (interfering with function); sensory loss or paresthesia interfering with ADLs (intefering with ADLs); permanent sensory loss that interferes with function (permanent sensory loss).
Time Frame: Baseline, Month 1, and Month 3
Population: as for outcome 8
Measure: Number; unit: participants
Arm/Group | Chemoradiation: Topotecan Plus WBRT | Radiation: WBRT Alone
Number analyzed (Participants) | 230 | 228
participants
  Baseline (BL), normal, n=230, 228 | 197 | 192
  Month (M) 1, normal, n=178, 180 | 144 | 159
  Month 3, normal, n=109, 107 | 100 | 94
  BL, not interfering with function, n=230, 228 | 26 | 26
  M 1, not interfering with function, n=178, 180 | 22 | 15
  M 3, not interfering with function, n=109, 107 | 5 | 9
  BL, interfering with function, n=230, 228 | 3 | 6
  M 1, interfering with function, n=178, 180 | 7 | 4
  M 3, interfering with function, n=109, 107 | 2 | 2
  Baseline, interfering with ADLs, n=230, 228 | 4 | 3
  Month 1, interfering with ADLs, n=178, 180 | 5 | 2
  Month 3, interfering with ADLs, n=109, 107 | 2 | 2
  Baseline, permanent sensory loss, n=230, 228 | 0 | 1

23. Secondary Outcome: Number of Participants With the Indicated Investigator Assessment of Ataxia (Right Upper Extremity: Finger to Nose Testing) at Baseline, Month 1, and Month 3
Description: The investigator assessed participants' status of ataxia (right upper extremity: finger to nose testing) and assigned each participant to one of the following categories: normal; Grade 1, asymptomatic but abnormal on physical examination, and not interfering with function; Grade 2, mild symptoms interfering with function, but not interfering with ADLs; Grade 3, moderate symptoms interfering with ADLs; Grade 4, bedridden or disabling.
Time Frame: Baseline, Month 1, and Month 3
Population: as for outcome 8
Measure: Number; unit: participants
Arm/Group | Chemoradiation: Topotecan Plus WBRT | Radiation: WBRT Alone
Number analyzed (Participants) | 229 | 228
participants
  Baseline, normal, n=229, 228 | 206 | 198
  Month 1, normal, 178, 179 | 166 | 166
  Month 3, normal, n=109, 107 | 103 | 95
  Baseline, Grade 1, n=229, 228 | 13 | 17
  Month 1, Grade 1, 178, 179 | 7 | 6
  Month 3, Grade 1, n=109, 107 | 6 | 5
  Baseline, Grade 2, n=229, 228 | 5 | 12
  Month 1, Grade 2, 178, 179 | 3 | 6
  Month 3, Grade 2, n=109, 107 | 0 | 5
  Baseline, Grade 3, n=229, 228 | 3 | 1
  Month 3, Grade 3, n=109, 107 | 0 | 1
  Baseline, Grade 4, n=229, 228 | 2 | 0
  Month 1, Grade 4, 178, 179 | 2 | 1
  Month 3, Grade 4, n=109, 107 | 0 | 1

24. Secondary Outcome: Number of Participants With the Indicated Investigator Assessment of Ataxia (Left Upper Extremity: Finger to Nose Testing) at Baseline, Month 1, and Month 3
Description: The investigator assessed participants' status of ataxia (left upper extremity: finger to nose testing) and assigned each participant to one of the following categories: normal; Grade 1, asymptomatic but abnormal on physical examination, and not interfering with function; Grade 2, mild symptoms interfering with function, but not interfering with ADLs; Grade 3, moderate symptoms interfering with ADLs; Grade 4, bedridden or disabling.
Time Frame: Baseline, Month 1, and Month 3
Population: as for outcome 8
Measure: Number; unit: participants
Arm/Group | Chemoradiation: Topotecan Plus WBRT | Radiation: WBRT Alone
Number analyzed (Participants) | 230 | 227
participants
  Baseline, normal, n=230, 227 | 199 | 201
  Month 1, normal, n=178, 178 | 156 | 162
  Month 3, normal, n=109, 107 | 97 | 94
  Baseline, Grade 1, n=230, 227 | 15 | 13
  Month 1, Grade 1, n=178, 178 | 14 | 9
  Month 3, Grade 1, n=109, 107 | 10 | 6
  Baseline, Grade 2, n=230, 227 | 8 | 7
  Month 1, Grade 2, n=178, 178 | 6 | 3
  Month 3, Grade 2, n=109, 107 | 2 | 3
  Baseline, Grade 3, n=230, 227 | 8 | 4
  Month 1, Grade 3, n=178, 178 | 0 | 3
  Month 3, Grade 3, n=109, 107 | 0 | 1
  Baseline, Grade 4, n=230, 227 | 0 | 2
  Month 1, Grade 4, n=178, 178 | 2 | 1
  Month 3, Grade 4, n=109, 107 | 0 | 3

25. Secondary Outcome: Number of Participants With the Indicated Investigator Assessment of Ataxia (Gait) at Baseline, Month 1, and Month 3
Description: The investigator assessed participants' status of ataxia (gait) and assigned each participant to one of the following categories: normal; Grade 1, asymptomatic but abnormal on physical examination, and not interfering with function; Grade 2, mild symptoms interfering with function, but not interfering with ADLs; Grade 3, moderate symptoms interfering with ADLs; Grade 4, bedridden or disabling.
Time Frame: Baseline, Month 1, and Month 3
Population: as for outcome 8
Measure: Number; unit: participants
Arm/Group | Chemoradiation: Topotecan Plus WBRT | Radiation: WBRT Alone
Number analyzed (Participants) | 230 | 227
participants
  Baseline, normal, n=230, 227 | 172 | 178
  Month 1, normal, n=178, 179 | 138 | 147
  Month 3, normal, n=108, 107 | 85 | 76
  Baseline, Grade 1, n=230, 227 | 13 | 22
  Month 1, Grade 1, n=178, 179 | 16 | 13
  Month 3, Grade 1, n=108, 107 | 9 | 10
  Baseline, Grade 2, n=230, 227 | 37 | 20
  Month 1, Grade 2, n=178, 179 | 14 | 14
  Month 3, Grade 2, n=108, 107 | 9 | 12
  Baseline, Grade 3, n=230, 227 | 6 | 6
  Month 1, Grade 3, n=178, 179 | 7 | 3
  Month 3, Grade 3, n=108, 107 | 4 | 5
  Baseline, Grade 4, n=230, 227 | 2 | 1
  Month 1, Grade 4, n=178, 179 | 3 | 2
  Month 3, Grade 4, n=108, 107 | 1 | 4

26. Secondary Outcome: Number of Participants With the Indicated Investigator Assessment of Ataxia (Balance) at Baseline, Month 1, and Month 3
Description: The investigator assessed participants' status of ataxia (balance) and assigned each participant to one of the following categories: normal; Grade 1, asymptomatic but abnormal on physical examination, and not interfering with function; Grade 2, mild symptoms interfering with function, but not interfering with ADLs; Grade 3, moderate symptoms interfering with ADLs; Grade 4, bedridden or disabling.
Time Frame: Baseline, Month 1, and Month 3
Population: as for outcome 8
Measure: Number; unit: participants
Arm/Group | Chemoradiation: Topotecan Plus WBRT | Radiation: WBRT Alone
Number analyzed (Participants) | 230 | 228
participants
  Baseline, normal, n=230, 228 | 153 | 152
  Month 1, normal, n=178, 178 | 131 | 128
  Month 3, normal, n=108, 107 | 78 | 75
  Baseline, Grade 1, n=230, 228 | 37 | 44
  Month 1, Grade 1, n=178, 178 | 23 | 28
  Month 3, Grade 1, n=108, 107 | 17 | 13
  Baseline, Grade 2, n=230, 228 | 27 | 23
  Month 1, Grade 2, n=178, 178 | 13 | 16
  Month 3, Grade 2, n=108, 107 | 8 | 9
  Baseline, Grade 3, n=230, 228 | 10 | 7
  Month 1, Grade 3, n=178, 178 | 8 | 5
  Month 3, Grade 3, n=108, 107 | 4 | 5
  Baseline, Grade 4, n=230, 228 | 3 | 2
  Month 1, Grade 4, n=178, 178 | 3 | 1
  Month 3, Grade 4, n=108, 107 | 1 | 5

27. Secondary Outcome: Number of Participants With Any Adverse Event (AE; Both Serious and Non-serious) or Serious Adverse Event (SAE)
Description: An AE is defined as any untoward medical occurrence in a patient or clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose: results in death; is life threatening; requires hospitalization or prolongation of existing hospitalization; results in disability/incapacity; is a congenital anomaly/birth defect. For a list of all SAEs and AEs, see the SAE/AE module of this results summary.
Time Frame: From Randomization until the last clinic visit associated with the study, up until 35 days after the start of the last course of treatment (up to 75 weeks)
Population: Modified ITT Population: all randomized participants who received at least one dose of randomized therapy. Participants were analyzed by the actual treatment received, even if this differed from the treatment to which they were randomized.
Measure: Number; unit: participants
Arm/Group | Chemoradiation: Topotecan Plus WBRT | Radiation: WBRT Alone
Number analyzed (Participants) | 235 | 233
participants
  AE | 204 | 148
  SAE | 96 | 43

28. Secondary Outcome: Number of Participants With the Indicated Worst-case Change From Baseline in the Indicated Chemistry Parameters With Respect to the Normal Range
Description: The worst-case change from Baseline in chemistry parameters was measured as decrease to low (DTL), change to normal or no change (CTN/NC), or increase to high (ITH). The worst-case change value could have been measured at any point during the on-therapy period. Participants are counted twice if the participant "Decreased to Low" and "Increased to High" during the on-therapy period.
Time Frame: as for outcome 27
Population: Modified ITT Population. Only those participants with available laboratory values (indicated by the "n" in the category titles) were analyzed. Different participants may have been analyzed for different parameters; therefore, the overall number of participants analyzed reflects everyone in the Modified ITT Population.
Measure: Number; unit: participants
Arm/Group | Chemoradiation: Topotecan Plus WBRT | Radiation: WBRT Alone
Number analyzed (Participants) | 235 | 233
participants
  Chloride, DTL, n=169, 171 | 32 | 21
  Chloride, CTN/NC, n=169, 171 | 116 | 144
  Chloride, ITH, n=169, 171 | 22 | 6
  Creatinine clearance, DTL, n=159, 145 | 26 | 9
  Creatinine clearance, CTN/NC, n=159, 145 | 121 | 134
  Creatinine clearance, ITH, n=159, 145 | 15 | 2
  Lactate dehydrogenase, DTL, n=169, 168 | 8 | 1
  Lactate dehydrogenase, CTN/NC, n=169, 168 | 117 | 127
  Lactate dehydrogenase, ITH, n=169, 168 | 47 | 40
  Total protein, DTL, n=171, 175 | 48 | 36
  Total protein, CTN/NC, n=171, 175 | 119 | 137
  Total protein, ITH, n=171, 175 | 4 | 2
  Urea/blood urea nitrogen, DTL, n=178, 179 | 7 | 4
  Urea/blood urea nitrogen, CTN/NC, n=178, 179 | 139 | 152
  Urea/blood urea nitrogen, ITH, n=178, 179 | 33 | 24
  Uric acid, DTL, n=159, 152 | 21 | 12
  Uric acid, CTN/NC, n=159, 152 | 125 | 134
  Uric acid, ITH, n=159, 152 | 13 | 6
  Basophils, DTL, n=215, 211 | 7 | 1
  Basophils, CTN/NC, n=215, 211 | 186 | 200
  Basophils, ITH, n=215, 211 | 25 | 10
  Eosinophils, DTL, n=214, 211 | 28 | 12
  Eosinophils, CTN/NC, n=214, 211 | 182 | 191
  Eosinophils, ITH, n=214, 211 | 4 | 8
  Hematocrit, DTL, n=215, 212 | 98 | 38
  Hematocrit, CTN/NC, n=215, 212 | 117 | 169
  Hematocrit, ITH, n=215, 212 | 1 | 6
  Monocytes, DTL, n=216, 212 | 84 | 17
  Monocytes, CTN/NC, n=216, 212 | 119 | 161
  Monocytes, ITH, n=216, 212 | 54 | 37
  Red Blood Cell Count, DTL, n=216, 212 | 103 | 38
  Red Blood Cell Count, CTN/NC, n=216, 212 | 113 | 171
  Red Blood Cell Count, ITH, n=216, 212 | 0 | 4

29. Secondary Outcome: Lesion Assessment and Measurement
Description: Lesions were assessed per WHO criteria. For lesion assessment data, see the outcome measure entitled "Number of participants with a complete response (CR) or a partial response (PR) (central nervous system [CNS]-radiologic)."
Time Frame: From the time of Randomization until the time of CR or PR (up to 75 weeks)
Arm/Group | Chemoradiation: Topotecan Plus WBRT | Radiation: WBRT Alone
Number analyzed (Participants) | 0 | 0

30. Secondary Outcome: Brain Symptoms
Description: Brain symptoms were assessed as the number of participants with neurological signs and symptoms. For brain symptom data, see the outcome measures entitled "Number of participants with the indicated investigator assessment for the neurological sign and symptom of X at Baseline, Month 1, and Month 3."
Time Frame: Baseline, Month 1, and Month 3
Arm/Group | Chemoradiation: Topotecan Plus WBRT | Radiation: WBRT Alone
Number analyzed (Participants) | 0 | 0

31. Secondary Outcome: Number of Participants Who Died or Progressed
Description: Disease-related events were measured as the number of participants who died or progressed. Progressive disease (PD) is defined as an increase >=25% in any measurable lesion or, in participants with non-measurable disease only, an estimation of an increase >=25%. In both cases, determination of progression included the appearance of any new lesions, or signification worsening of conditions presumed to be related to malignancy. Participants with clinical or laboratory evidence of possible disease progression were to be evaluated radiologically. Data were analyzed with censoring for extended loss to follow-up to account for two or more missed assessments before an event. The date of the last adequate CNS assessment before extended loss to follow-up was used for censored participants.
Time Frame: as for outcome 27
Population: mITT Population
Measure: Number; unit: participants
Arm/Group | Chemoradiation: Topotecan Plus WBRT | Radiation: WBRT Alone
Number analyzed (Participants) | 235 | 233
participants | 179 | 161

ADVERSE EVENTS:
Description: Serious adverse events (SAEs) and non-serious AEs were collected in members of the Modified Intent-to-Treat Population, comprised of all randomized participants (par.) who received at least one dose of randomized therapy. Par. were analyzed by the actual treatment received, even if it differed from the treatment to which they were randomized.
Arm/Group | Chemoradiation: Topotecan Plus WBRT | Radiation: WBRT Alone
Serious Adverse Events (participants affected / at risk) | 96/235 | 43/233
Other Adverse Events (participants affected / at risk) | 192/235 | 139/233
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Chemoradiation: Topotecan Plus WBRT (N=235) | Radiation: WBRT Alone (N=233)
Neutropenia (Blood and lymphatic system disorders) | 22 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 22 | 1
Anaemia (Blood and lymphatic system disorders) | 16 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 13 | 0
Pneumonia (Infections and infestations) | 7 | 6
Leukopenia (Blood and lymphatic system disorders) | 8 | 1
Dehydration (Metabolism and nutrition disorders) | 5 | 3
Asthenia (General disorders) | 5 | 1
Diarrhoea (Gastrointestinal disorders) | 6 | 0
Pancytopenia (Blood and lymphatic system disorders) | 6 | 0
Pyrexia (General disorders) | 5 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Sepsis (Infections and infestations) | 4 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Deep vein thrombosis (Vascular disorders) | 3 | 1
Dyspnoea (Gastrointestinal disorders) | 3 | 1
Brain oedema (Nervous system disorders) | 3 | 0
Disease progression (General disorders) | 3 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 3 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Septic shock (Infections and infestations) | 1 | 2
Vomiting (Gastrointestinal disorders) | 3 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 2 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 1
Cardiac failure acute (Cardiac disorders) | 2 | 0
Cerebrovascular accident (Nervous system disorders) | 2 | 0
Confusional state (Psychiatric disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 0 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 1
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Overdose (Injury, poisoning and procedural complications) | 2 | 0
Performance status decreased (General disorders) | 2 | 0
Pericarditis (Cardiac disorders) | 1 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Small intestinal haemorrhage (Gastrointestinal disorders) | 2 | 0
Syncope (Nervous system disorders) | 2 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 1 | 0
Agranulocytosis (Blood and lymphatic system disorders) | 1 | 0
Arterial thrombosis limb (Vascular disorders) | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Blood bilirubin increased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Cardiopulmonary failure (Cardiac disorders) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Convulsion (Nervous system disorders) | 1 | 0
Coronary artery insufficiency (Cardiac disorders) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 1
Encephalopathy (Nervous system disorders) | 1 | 0
Face injury (Injury, poisoning and procedural complications) | 1 | 0
Fatigue (General disorders) | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
General physical health deterioration (General disorders) | 1 | 0
Grand mal convulsion (Nervous system disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0
Hydrocephalus (Nervous system disorders) | 1 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Intestinal perforation (Gastrointestinal disorders) | 1 | 0
Jugular vein thrombosis (Vascular disorders) | 1 | 0
Lobar pneumonia (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Lung abscess (Infections and infestations) | 1 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 0 | 1
Oesophageal stenosis (Gastrointestinal disorders) | 0 | 1
Oropharyngeal pain (Gastrointestinal disorders) | 1 | 0
Oropharyngitis fungal (Infections and infestations) | 1 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0
Pain (General disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Paraplegia (Nervous system disorders) | 1 | 0
Peridiverticular abscess (Infections and infestations) | 1 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Radiation pneumonitis (Injury, poisoning and procedural complications) | 0 | 1
Radiculopathy (Nervous system disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 1
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 0 | 1
Superior vena cava syndrome (Vascular disorders) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1
Venous thrombosis (Vascular disorders) | 0 | 1
Weight decreased (Investigations) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Chemoradiation: Topotecan Plus WBRT (N=235) | Radiation: WBRT Alone (N=233)
Nausea (Gastrointestinal disorders) | 64 | 30
Vomiting (Gastrointestinal disorders) | 37 | 24
Diarrhoea (Gastrointestinal disorders) | 19 | 8
Dyspepsia (Gastrointestinal disorders) | 17 | 10
Constipation (Gastrointestinal disorders) | 8 | 10
Abdominal pain (Gastrointestinal disorders) | 4 | 6
Stomatitis (Gastrointestinal disorders) | 7 | 1
Abdominal pain upper (Gastrointestinal disorders) | 2 | 3
Dysphagia (Gastrointestinal disorders) | 2 | 3
Dry mouth (Gastrointestinal disorders) | 2 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 1
Flatulence (Gastrointestinal disorders) | 2 | 0
Mouth ulceration (Gastrointestinal disorders) | 2 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 1
Breath odour (Gastrointestinal disorders) | 0 | 1
Faecal incontinence (Gastrointestinal disorders) | 1 | 0
Faeces discoloured (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1
Gingival pain (Gastrointestinal disorders) | 1 | 0
Glossodynia (Gastrointestinal disorders) | 1 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Hyperchlorhydria (Gastrointestinal disorders) | 1 | 0
Oesophageal pain (Gastrointestinal disorders) | 1 | 0
Oral pain (Gastrointestinal disorders) | 0 | 1
Retching (Gastrointestinal disorders) | 1 | 0
Fatigue (General disorders) | 39 | 37
Asthenia (General disorders) | 29 | 19
Oedema peripheral (General disorders) | 15 | 15
Pyrexia (General disorders) | 13 | 5
Mucosal inflammation (General disorders) | 7 | 0
Gait disturbance (General disorders) | 2 | 4
Face oedema (General disorders) | 1 | 3
Pain (General disorders) | 1 | 3
Chest pain (General disorders) | 1 | 2
Chills (General disorders) | 2 | 1
Non-cardiac chest pain (General disorders) | 2 | 1
Spinal pain (General disorders) | 1 | 1
Chest discomfort (General disorders) | 0 | 1
Early satiety (General disorders) | 1 | 0
Gravitational oedema (General disorders) | 1 | 0
Hyperthermia (General disorders) | 0 | 1
Influenza like illness (General disorders) | 1 | 0
Local swelling (General disorders) | 0 | 1
Localised oedema (General disorders) | 0 | 1
Malaise (General disorders) | 1 | 0
Mucosal erosion (General disorders) | 1 | 0
Oedema (General disorders) | 1 | 0
Swelling (General disorders) | 1 | 0
Headache (Nervous system disorders) | 27 | 28
Dizziness (Nervous system disorders) | 27 | 19
Somnolence (Nervous system disorders) | 14 | 14
Hypoaesthesia (Nervous system disorders) | 6 | 11
Ataxia (Nervous system disorders) | 8 | 6
Coordination abnormal (Nervous system disorders) | 7 | 4
Tremor (Nervous system disorders) | 6 | 4
Paraesthesia (Nervous system disorders) | 5 | 4
Amnesia (Nervous system disorders) | 2 | 6
Dysgeusia (Nervous system disorders) | 6 | 2
Aphasia (Nervous system disorders) | 1 | 6
Balance disorder (Nervous system disorders) | 0 | 7
Convulsion (Nervous system disorders) | 4 | 1
Epilepsy (Nervous system disorders) | 1 | 3
Neuropathy peripheral (Nervous system disorders) | 2 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 2 | 2
Speech disorder (Nervous system disorders) | 1 | 3
Syncope (Nervous system disorders) | 2 | 1
Brain oedema (Nervous system disorders) | 1 | 1
Convulsions local (Nervous system disorders) | 2 | 0
Hemiparesis (Nervous system disorders) | 0 | 2
Hemiplegia (Nervous system disorders) | 1 | 1
Loss of consciousness (Nervous system disorders) | 1 | 1
Memory impairment (Nervous system disorders) | 1 | 1
Psychomotor hyperactivity (Nervous system disorders) | 0 | 2
Ageusia (Nervous system disorders) | 0 | 1
Alcoholic seizure (Nervous system disorders) | 0 | 1
Burning sensation (Nervous system disorders) | 1 | 0
Cognitive disorder (Nervous system disorders) | 1 | 0
Dysarthria (Nervous system disorders) | 0 | 1
Facial paresis (Nervous system disorders) | 1 | 0
Hypersomnia (Nervous system disorders) | 0 | 1
Hypotonia (Nervous system disorders) | 1 | 0
Mental impairment (Nervous system disorders) | 0 | 1
Monoplegia (Nervous system disorders) | 1 | 0
Neuritis (Nervous system disorders) | 0 | 1
Paresis (Nervous system disorders) | 1 | 0
Partial seizures (Nervous system disorders) | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0
Polyneuropathy (Nervous system disorders) | 0 | 1
Sciatica (Nervous system disorders) | 0 | 1
Visual field defect (Nervous system disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 31 | 20
Cough (Respiratory, thoracic and mediastinal disorders) | 26 | 17
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 | 7
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Hiccups (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 29 | 22
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 2
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Extremity contracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 28 | 17
Increased appetite (Metabolism and nutrition disorders) | 7 | 6
Hypokalaemia (Metabolism and nutrition disorders) | 9 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 4 | 3
Dehydration (Metabolism and nutrition disorders) | 2 | 4
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 1
Cachexia (Metabolism and nutrition disorders) | 2 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 1 | 0
Polydipsia (Metabolism and nutrition disorders) | 1 | 0
Pneumonia (Infections and infestations) | 4 | 4
Oral candidiasis (Infections and infestations) | 5 | 2
Urinary tract infection (Infections and infestations) | 3 | 4
Candidiasis (Infections and infestations) | 3 | 2
Oral fungal infection (Infections and infestations) | 2 | 3
Oropharyngitis fungal (Infections and infestations) | 1 | 3
Upper respiratory tract infection (Infections and infestations) | 3 | 1
Nasopharyngitis (Infections and infestations) | 1 | 2
Rhinitis (Infections and infestations) | 2 | 1
Bronchitis (Infections and infestations) | 0 | 2
Cystitis (Infections and infestations) | 0 | 2
Herpes zoster (Infections and infestations) | 0 | 2
Influenza (Infections and infestations) | 2 | 0
Oesophageal candidiasis (Infections and infestations) | 2 | 0
Oral herpes (Infections and infestations) | 2 | 0
Oropharyngeal candidiasis (Infections and infestations) | 2 | 0
Pharyngitis (Infections and infestations) | 2 | 0
Anal fungal infection (Infections and infestations) | 1 | 0
Fungal infection (Infections and infestations) | 0 | 1
Fungal oesophagitis (Infections and infestations) | 0 | 1
Furuncle (Infections and infestations) | 0 | 1
Herpes simplex (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 0 | 1
Mastoiditis (Infections and infestations) | 0 | 1
Orchitis (Infections and infestations) | 0 | 1
Otitis media (Infections and infestations) | 0 | 1
Rash pustular (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1
Soft tissue infection (Infections and infestations) | 1 | 0
Tonsillitis (Infections and infestations) | 1 | 0
Tracheobronchitis (Infections and infestations) | 0 | 1
Vaginal infection (Infections and infestations) | 1 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 1 | 0
Insomnia (Psychiatric disorders) | 17 | 19
Confusional state (Psychiatric disorders) | 7 | 11
Anxiety (Psychiatric disorders) | 4 | 1
Depression (Psychiatric disorders) | 2 | 2
Mood altered (Psychiatric disorders) | 0 | 2
Nervousness (Psychiatric disorders) | 0 | 2
Delusion (Psychiatric disorders) | 0 | 1
Depressed mood (Psychiatric disorders) | 1 | 0
Disorientation (Psychiatric disorders) | 0 | 1
Initial insomnia (Psychiatric disorders) | 0 | 1
Mental disorder (Psychiatric disorders) | 1 | 0
Sleep disorder (Psychiatric disorders) | 0 | 1
Staring (Psychiatric disorders) | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 21 | 17
Erythema (Skin and subcutaneous tissue disorders) | 4 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 3
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 2
Swelling face (Skin and subcutaneous tissue disorders) | 1 | 2
Acne (Skin and subcutaneous tissue disorders) | 1 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 1
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 2
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 1 | 0
Increased tendency to bruise (Skin and subcutaneous tissue disorders) | 0 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 1
Weight decreased (Investigations) | 18 | 8
Blood lactate dehydrogenase increased (Investigations) | 3 | 2
Platelet count decreased (Investigations) | 4 | 1
Haemoglobin decreased (Investigations) | 3 | 1
Alanine aminotransferase increased (Investigations) | 2 | 1
Weight increased (Investigations) | 2 | 1
Blood glucose increased (Investigations) | 0 | 2
Neutrophil count decreased (Investigations) | 2 | 0
White blood cell count decreased (Investigations) | 1 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Bacterial test positive (Investigations) | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 1
Blood creatinine increased (Investigations) | 0 | 1
Blood magnesium increased (Investigations) | 1 | 0
Blood phosphorus decreased (Investigations) | 0 | 1
Blood phosphorus increased (Investigations) | 1 | 0
Blood urea increased (Investigations) | 0 | 1
Blood uric acid increased (Investigations) | 0 | 1
Body temperature increased (Investigations) | 1 | 0
Breath sounds abnormal (Investigations) | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 1
International normalised ratio increased (Investigations) | 1 | 0
Vision blurred (Eye disorders) | 4 | 8
Visual acuity reduced (Eye disorders) | 3 | 2
Visual impairment (Eye disorders) | 2 | 2
Asthenopia (Eye disorders) | 1 | 0
Blindness (Eye disorders) | 0 | 1
Conjunctivitis (Eye disorders) | 0 | 1
Eye inflammation (Eye disorders) | 1 | 0
Eye pain (Eye disorders) | 1 | 0
Myopia (Eye disorders) | 1 | 0
Retinal vascular disorder (Eye disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 4 | 3
Tinnitus (Ear and labyrinth disorders) | 4 | 0
Ear pain (Ear and labyrinth disorders) | 2 | 0
Ear pruritus (Ear and labyrinth disorders) | 2 | 0
Auricular swelling (Ear and labyrinth disorders) | 0 | 1
Deafness (Ear and labyrinth disorders) | 0 | 1
Hearing impaired (Ear and labyrinth disorders) | 1 | 0
Hypoacusis (Ear and labyrinth disorders) | 1 | 0
Hypotension (Vascular disorders) | 6 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 2
Hypertension (Vascular disorders) | 2 | 1
Flushing (Vascular disorders) | 1 | 1
Phlebitis (Vascular disorders) | 2 | 0
Haematoma (Vascular disorders) | 0 | 1
Hot flush (Vascular disorders) | 0 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 1
Thrombophlebitis superficial (Vascular disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 7 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 5 | 1
Neutropenia (Blood and lymphatic system disorders) | 3 | 0
Leukopenia (Blood and lymphatic system disorders) | 2 | 0
Coagulopathy (Blood and lymphatic system disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 3 | 2
Tachycardia (Cardiac disorders) | 2 | 3
Cardiac failure (Cardiac disorders) | 1 | 1
Palpitations (Cardiac disorders) | 2 | 0
Angina pectoris (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 1
Supraventricular extrasystoles (Cardiac disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 2 | 1
Dysuria (Renal and urinary disorders) | 2 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 1
Chromaturia (Renal and urinary disorders) | 0 | 1
Incontinence (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1
Urinary bladder haemorrhage (Renal and urinary disorders) | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 3
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 1
Thermal burn (Injury, poisoning and procedural complications) | 1 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Incision site pain (Injury, poisoning and procedural complications) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 1
Radiation skin injury (Injury, poisoning and procedural complications) | 1 | 0
Skin wound (Injury, poisoning and procedural complications) | 1 | 0
Cushingoid (Endocrine disorders) | 1 | 1
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 | 0
Epididymitis (Reproductive system and breast disorders) | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.